CLINICAL TRIAL: NCT04912830
Title: Tension Free Vaginal Tape Surgery - Follow up After 10 and 20 Years: Success Rate and Long-term Complications
Brief Title: Tension Free Vaginal Tape Surgery - Follow up After 10 and 20 Years
Acronym: TVTOPP
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Alesund Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 141799
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Urinary Incontinence,Stress
Keywords: Surgery; Suburethral Slings; Tension-free vaginal tape
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Suburethral Slings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 20 years follow-up after TVT surgery: Women who had tension free vaginal tape surgery during January 2001-December 2002 in Norway, identified in the National Incontinence Registry
  Interventions: Procedure: Tension-free vaginal tape
- 10 years follow-up after TVT surgery, age 42 or younger: Women who had tension free vaginal tape surgery and aged < 42 years at the time of surgery during 2011-2012 in Norway, identified in the National Incontinence Registry
  Interventions: Procedure: Tension-free vaginal tape

INTERVENTIONS:
Procedure: Tension-free vaginal tape — female incontinence surgery with polypropylene tape applied

SUMMARY:
Over the past 5-7 years there has been increasing concern about the use of polypropylene tapes in female incontinence surgery. There has been a special focus on pain in the vagina and lower abdomen and pain during sexual intercourse. Some have also asked if the polypropylene tape could cause impairment of the immune system leading to allergy, connective tissue disorders etc. There are still only a few publications on complications after sling surgery.

In Norway it is mandatory to register all incontinence surgery in the National incontinence registry (Norsk Kvinnelig Inkontinens Register (NKIR). In 2019 >99 % of all procedures were registered in this registry. Data about type and severity of incontinence are registered, as well as complications at surgery. The same data are entered at a 6 months and 3 years follow up. Data for the follow up visits are not complete. The NKIR registry and other similar registries have been criticized for not following the women long enough and therefore missing important information regarding long-term complications. Few studies have followed the women for a longer time after surgery. The main aim of this study is to find the prevalence of women still satisfied with the TVT surgery and the prevalence of long-term complications after 10 and 20 years.

ELIGIBILITY:
Inclusion Criteria:

* had TVT surgery in Norway January 2001-December 2002 (20-years follow-up cohort)
* had TVT surgery in Norway, < 42 years at the time of surgery in 2011-2012 (10-years follow-up cohort)

Exclusion Criteria:

* Dead
* Not willing to participate
* Moved out of Norway

Ages: 40 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who had tension free vaginal tape surgery 10 and 20 years ago in Norway, identified in the National Incontinence Registry (Norsk Kvinnelig Inkontinens Register (NKIR).
Sampling Method: Non-Probability Sample
Enrollment: 1210 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
prevalence of persistant pelvic pain after TVT surgery | 20 years
prevalence or persistant pelvic pain after TVT surgery | 10 years
subjective cure rate | 20 years
  assessed by stress index; stress index <=3 is considered 'successful'
subjective cure rate | 10 years
  assessed by stress index; stress index <=3 is considered 'successful'
Urinary bladder microbiota | 20 years
  assessed by quadruplex PCR
Urinary bladder microbiota | 10 years
  assessed by quadruplex PCR
Tension free vaginal tape placement along the urethra assessed with ultrasound | 20 years
Tension free vaginal tape placement along the urethra assessed with ultrasound | 10 years
Sexually active | 20 years
  yes/no question
Sexually active | 10 years
  yes/no question
Levator avulsion assessed by ultrasound | 20 years
Levator avulsion assessed by ultrasound | 10 years

SECONDARY OUTCOMES:
prevalence of surgical TVT removal | 20 years
prevalence of surgical TVT removal | 10 years
Prevalence of recurrent surgery for stress urinary incontinence | 20 years
prevalence of recurrent surgery for stress urinary incontinence | 10 years
Quality of life assessed by RAND-36 questionnaire | 20 years
  The RAND 36-Item Health Survey 1.0 (distributed by RAND, Norwegian translation)
Quality of life assessed by RAND-36 questionnaire | 10 years
  The RAND 36-Item Health Survey 1.0 (distributed by RAND, Norwegian translation)
Pelvic organ prolapse assessed by POP-Q at clinical examination | 20 years
  Pelvic organ prolapse quantification system (POP-Q)
Pelvic organ prolapse assessed by POP-Q at clinical examination | 10 years
  Pelvic organ prolapse quantification system (POP-Q)
Symptoms of pelvic floor disorders assessed by PFDI questionnaire | 20 years
  Pelvic floor distress inventory (PFDI)
Symptoms of pelvic floor disorders assessed by PFDI questionnaire | 10 years
  Pelvic floor distress inventory (PFDI)

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Baade Rø, phd prof, Study Director — NTNU, Department of Clinical and Molecular Medicine
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solhaug BR, Svenningsen R, Nyhus MO, Volloyhaug I. Long-term sexual function after mid-urethral slings for stress urinary incontinence in women. Acta Obstet Gynecol Scand. 2024 Aug;103(8):1664-1671. doi: 10.1111/aogs.14894. Epub 2024 Jun 13. PMID 38867580